CLINICAL TRIAL: NCT06708598
Title: Learning Curve of Ultrasound-Guided Suprainguinal Fascia Iliaca Block: A Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Senay Canikli (Other)
Responsible Party: Sponsor-Investigator, Senay Canikli, MD, Samsun University
Organization: Samsun University (Other)
Other Study IDs: GOKAEK 2024/21/6
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Learning Curve; Suprainguinal Fasya Iliaca Block; Ultrasound-guided Regional Anesthesia (UGRA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Competence in ultrasound-guided regional anesthesia (UGRA) requires practitioners to acquire cognitive and technical skills. Various difficulties have been identified in anesthesia residents' learning UGRA skills. There is currently no approved UGRA curriculum for residents, and the level of UGRA proficiency achieved during residency may vary significantly. However, no specific training criteria have been defined for this block. It is important to establish criteria to evaluate the adequacy of education.

DETAILED DESCRIPTION:
Compared to other nerve localization techniques, the benefits of UGRA include higher nerve block success rates, faster onset times, reduced local anesthetic volumes, and a lower risk of local anesthetic-related complications. Most experts now consider ultrasound guidance as the standard of care for peripheral nerve blocks. Successfully performing a UGRA procedure requires a triad of three distinct but interrelated skills: image acquisition, anatomical interpretation, and hand-eye coordination.

In our clinic, we routinely perform various nerve block techniques under ultrasound guidance during the perioperative period, both for postoperative analgesia and as a primary anesthetic method. Specifically, in our clinic, the suprainguinal fascia iliaca block (SIFIB) is routinely applied for postoperative analgesia, particularly in orthopedic cases. Before performing a nerve block procedure, resident doctors in our clinic undergo standard training and subsequently perform blocks under the supervision and support of experienced specialists and academicians.

ELIGIBILITY:
Inclusion Criteria:

- Anesthesia residents with less than 2 years of anesthesia experience who have never performed a SIFIB before

Exclusion Criteria:

* Having previously performed a SIFIB

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Anesthesia residents with less than 2 years of anesthesia experience who have never performed a SIFIB before.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Block success | 20 minute
  "Additionally, to evaluate the success of the procedure more objectively, the following parameters will be assessed using a 5-point Likert scale (1: Very low, 2: Low, 3: Moderate, 4: High, 5: Very high). For the procedure to be considered successful, a score of 4 must be obtained for each parameter. These parameters include:
  * Placement of the ultrasound probe
  * Visualization of anatomical structures (muscle, bone, fascia, vessels)
  * Optimization of needle localization
  * Spread of the drug beneath the iliac fascia"

SECONDARY OUTCOMES:
Block performance time | 20 minute
  The block performance times of each practitioner will be recorded, and the average performance time will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Senay Canikli Adıgüzel, Study Director — Samsun University
Locations (1):
- SAMSUN UNIVERSITY Samsun Training and research hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study data can be shared upon appropriate request after the study is completed.

REFERENCES:
- [Background] Dang D, Kamal M, Kumar M, Paliwal B, Nayyar A, Bhatia P, Singariya G. Comparison of human cadaver and blue phantom for teaching ultrasound-guided regional anesthesia to novice postgraduate students of anesthesiology: A randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2024 Apr-Jun;40(2):276-282. doi: 10.4103/joacp.joacp_234_22. Epub 2024 May 16. PMID 38919433
- [Background] Kim TE, Tsui BCH. Simulation-based ultrasound-guided regional anesthesia curriculum for anesthesiology residents. Korean J Anesthesiol. 2019 Feb;72(1):13-23. doi: 10.4097/kja.d.18.00317. Epub 2018 Nov 27. PMID 30481945
- [Background] Rossetti M, Allgower D, Hell K. [Azygoportal interruption, fundoplication and vagotomy in hemorrhagic esophageal varices]. Helv Chir Acta. 1977 Oct;44(4):481-4. German. PMID 309462